CLINICAL TRIAL: NCT06785324
Title: Nutrition and Exercise to Optimize Muscle and Adiposity in Adults With ALL: NEOMA ALL Trial
Brief Title: Study of Nutrition and Exercise in Adults Hospitalized for Treatment of Acute Lymphoblastic Leukemia (ALL)
Acronym: NEOMA ALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB24-1500
Record Dates: First submitted 2024-12-23; First posted 2025-01-21 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Philadelphia Chromosome Negative; B Cell Acute Lymphoblastic Leukemia (B-ALL); B-ALL
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nutrition and Exercise interventions (Experimental): Participants will receive an exercise and nutrition (diet) intervention while hospitalized for routine treatment for their ALL.
  Interventions: Behavioral: Nutrition Intervention; Behavioral: Exercise intervention

INTERVENTIONS:
Behavioral: Nutrition Intervention — The nutrition intervention will target a 10% caloric deficit calculated from each patient's Basal Metabolic Rate (WHO/Schofield) utilizing a high protein (>25%), low fat (<25%), low glycemic index/high fiber (45-55%) diet.
  The study registered dietician (RD) will meet with the patient on day of enrollment to go over the "menu" of dietary options and will re-assess the patient every two days (excluding weekends) for adherence.
  My Plate (USDA) will control portion size and eating habits.
Behavioral: Exercise intervention — The exercise intervention will target 200 minutes of "moderate" physical activity weekly, as defined by Metabolic Equivalents (METs) of 3-6, made up of aerobic and resistance training activities tailored to the patient's preference by working with the study physical therapist (PT).
  Physical Therapist to evaluate patient every 48 hours, excluding weekends.

SUMMARY:
This clinical trial aims to assess the effect of nutrition and exercise on muscle and adiposity in adults with Philadelphia Chromosome (Ph) Negative B-ALL undergoing inpatient induction therapy.

Participants will take part in 2 different interventions:

* Nutrition Intervention
* Physical Exercise Intervention

All subjects will be provided with a wearable electronic activity monitor (FitBit®) to assist in recording activity levels in minutes of activity.

ELIGIBILITY:
Inclusion Criteria:

* New Diagnosis of Philadelphia Chromosome Negative B-ALL
* Receiving intensive pediatric-inspired induction chemotherapy

Exclusion Criteria:

* BMI ≤18.5 kg/m2 at time of diagnosis
* Unable to comply with both the recommended diet and exercise regimen as deemed by the research or treatment team
* Pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-11-06 (Estimated); Study Completion 2027-11-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of nutrition and exercise intervention | End of study recruitment (approximately 1 year)
  Percentage of eligible patients that consent to trial.

SECONDARY OUTCOMES:
Adherence to dietary intervention | 22 days
  Percentage of participants that are "adherent", defined as >75% of the patient's dietary assessments consistent with the prescribed diet.
Adherence to exercise intervention | 22 days
  Percentage of participants able to meet the exercise goal in 2 out of 3 weeks of induction therapy or 66% of their weeks of inpatient admission if admitted for more than 3 weeks.
Usability of interventions | 22 days
  To assess intervention usability, a 10-item questionnaire, the System Usability Scale Questionnaire, will be administered to each patient postintervention. This instrument rates responses from "strongly agree" to "strongly disagree". A score >68 is considered of acceptable usability.
Body composition changes - Visceral Adiposity | 22 days
  Percent change in Visceral Adiposity from baseline to day 22 on study will be described. CT measurements of height-adjusted lumber adiposity area (VAT) are calculated from routine contrast and non-contrast CT scans of chest and abdomen
Body composition changes - Sarcopenia (SMI) | 22 days
  Percent change in sarcopenia score from baseline to day 22 on study will be described. Sarcopenia is loss of skeletal muscle mass and function associated with aging and will be calculated as mg/m2 measurements of skeletal muscle cross-sectional area, index, and radiation attenuation utilizing clinical computed tomography (CT) scans. The lower the value the worse the outcome.
Impact on minimal residual disease (MRD) | 22 days
  Number of participants that are MRD positive at end of induction therapy
Impact on Treatment toxicities | 22 days
  Number of participants that experience experience grade 3-4 hyperglycemia and hepatoxicity during induction. Adverse Events will be graded using Common Terminology Criteria for Adverse Events (CTCAE) v5 criteria.
Changes to the Host Metabolome | 22 days
  Assessment of changes to the host metabolome throughout the intervention on daily serum samples (excluding weekends and holidays) will be assess descriptively

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided